CLINICAL TRIAL: NCT04782310
Title: Effectiveness of Adding Duloxetine to Pregabalin in Treatment of Acute Postoperative and Prevention of Chronic Pain Following Thoracotomy Surgeries; Randomized Controlled Study
Brief Title: Duloxetine vs Pregabalin for Thoracotomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-386-2020
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Pregabalin (Experimental): Patients will receive oral Pregabalin 75mg two hour preoperatively, 12 hours postoperative and will continue for one week twice per day.
  Interventions: Drug: Pregabalin
- Group Duloxetine (Experimental): Patients will receive oral duloxetine 30mg two hour preoperatively …will be continued for one week once per day after breakfast .
  Interventions: Drug: Duloxetine
- Group Pregabalin& Duloxetine (Experimental): Patients will receive single dose of Pregabalin 75mg + duloxetine 30mg two hour preoperatively, 75mg pregabalin 12 hour postoperative and then will continue pregabalin twice per day +duloxetine once after breakfast for one week.
  Interventions: Drug: Pregabalin; Drug: Duloxetine

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 75mg two hour preoperatively, 12 hours postoperative and will continue for one week twice per day.
  Arms: Group Pregabalin; Group Pregabalin& Duloxetine
Drug: Duloxetine — Duloxetine 30mg two hour preoperatively …will be continued for one week once per day after breakfast .
  Arms: Group Duloxetine; Group Pregabalin& Duloxetine

SUMMARY:
This study investigates the effects of preoperative use of oral combination of duloxetine and Pregabalin in comparison with preoperative oral Pregabalin only in treatment of acute postoperative and prevention of chronic pain following thoracotomy surgeries.

DETAILED DESCRIPTION:
75 Patients, undergoing thoracotomy surgery will be randomly allocated into three equal groups, each (n=25 ), using computerized generated random tables: Group P: will receive oral Pregabalin 75mg two hour preoperatively, 12 hours postoperative and will continue for one week twice per day.

Group D:will receive oral duloxetine 30mg two hour preoperatively …will be continued for one week once per day after breakfast .

Group C: will receive single dose of Pregabalin 75mg + duloxetine 30mg two hour preoperatively, 75mg pregabalin 12 hour postoperative and then will continue pregabalin twice per day +duloxetine once after breakfast for one week.

The total amount of morphine consumption in the first 24 hours postoperatively, total amount of intraoperative fentanyl will be recorded, change in hemodynamics ((heart rate and mean arterial blood pressure), respiratory rate and oxygen saturation will be monitored and recorded at 0,2, 4, 8, 12 ,16 &24 hours and Visual analogue scale at 0, 2,4, 8, 12, 16 &24 hours postoperatively then at 3rd, 5th days, 4th week and12th week will be measured.

ELIGIBILITY:
Inclusion Criteria:

* ● Physical status ASA II, III.

  * Age ≥ 18 and ≤ 65 Years.
  * Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.
  * Cancer patients undergoing posterolateral thoracotomy incision for cancer lung, mesothelioma or metastatectomy from the lung.
  * Patient is able to provide a written informed consent.

Exclusion Criteria:

* ● Patients with Known sensitivity or contraindication to drug used in the study

  * History of psychological disorders and/or chronic pain.
  * Previous administration of antidepressants, anticonvulsants, or opioids before surgery.
  * Patient refusal.
  * Severe respiratory or cardiac disorders.
  * Advanced liver or kidney disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 24 hours postoperative
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Visual analogue scale | 12 weeks
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Total dose of intraoperative fentanyl. | 2 hours intraoperative
  The total dose of intraoperative fentanyle administration rather than the dose used in induction
Heart rate | 24 hours
  Heart rate will be measured preoperative as baseline value, intraoperative and postoperative
Mean arterial pressure | 24 hours postoperative
  Mean arterial blood pressure will be measured preoperative as baseline value, intraoperative and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, Principal Investigator — Cairo University
Locations (1):
- Bassant abdelhamid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altiparmak B, Guzel C, Gumus Demirbilek S. Comparison of Preoperative Administration of Pregabalin and Duloxetine on Cognitive Functions and Pain Management After Spinal Surgery: A Randomized, Double-blind, Placebo-controlled Study. Clin J Pain. 2018 Dec;34(12):1114-1120. doi: 10.1097/AJP.0000000000000640. PMID 30020088
- [Background] Gilron I, Chaparro LE, Tu D, Holden RR, Milev R, Towheed T, DuMerton-Shore D, Walker S. Combination of pregabalin with duloxetine for fibromyalgia: a randomized controlled trial. Pain. 2016 Jul;157(7):1532-40. doi: 10.1097/j.pain.0000000000000558. PMID 26982602